CLINICAL TRIAL: NCT02229058
Title: Phase II Study of Albumin Bound Paclitaxel Plus S-1 as the First Line Chemotherapy in Advanced or Recurrent Gastric Cancer
Brief Title: Albumin Bound Paclitaxel Plus S-1 as the First Line Chemotherapy in Advanced or Recurrent Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor of Medical Oncology,Vice-president of Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-SG
Record Dates: First submitted 2014-03-08; First posted 2014-08-29 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Albumin Bound Paclitaxel; S-1; First Line
MeSH Terms: conditions — Stomach Neoplasms | interventions — Albumin-Bound Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albumin Bound Paclitaxel plus S-1 (Experimental): Abraxane 120 mg/m2, D1,D8;S-1 40~60mg QD D1-D14,every 3 weeks until disease progress or intolerable toxicity.
  Interventions: Drug: Albumin Bound Paclitaxel; Drug: S-1

INTERVENTIONS:
Drug: Albumin Bound Paclitaxel — 120 mg/m2, D1,D8,every 3 weeks until disease progress or intolerable toxicity.
  Other Names: abraxane
Drug: S-1 — 40mg QD D1-D14,every 3 weeks,for BSA<1.25 m2, 50mg QD D1-D14,every 3 weeks,for BSA=1.25～1.5m2, 60mg QD D1-D14,every 3 weeks,for BSA>1.5m2,until disease progress or intolerable toxicity.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of s-1 plus Albumin Bound Paclitaxel as first-line therapy in the treatment of patients with advanced gastric cancer.

DETAILED DESCRIPTION:
As the first phase II clinical trial of fluoropyrimidines plus Nab-PTX in AGC patientsphase II trial, this study aimed to evaluate the efficacy and safety of S-1 plus Nab-PTX as a first-line treatment for patients with metastatic gastric cancer. All patients were orally treated with S-1 in doses of 40 mg (BSA<1.25 m2), 50 mg (1.25≤BSA<1.50 m2) and 60 mg (BSA≥1.50 m2) b.i.d. on days 1-14 in combination with Nab-PTX (240 mg/m2, divided on days 1 and 8, intravenously for 30 minutes) of each 21-day cycle. Treatment was planned for 6 cycles or until progression, unacceptable toxicity, or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach with inoperable locally advanced or recurrent and/or metastatic disease.
* Male or female.
* Age ≥ 18.
* No previous chemotherapy for advanced/metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study).
* Measurable disease, according to the Response Evaluation Criteria in Solid Tumours(RECIST)
* ECOG Performance status 0, 1 or 2
* Haematological, Biochemical and Organ Function: Neutrophil count >2.0 × 10 9/L, platelet count > 100 ×10 9/L. Serum bilirubin< 1.5 × upper limit of normal (ULN); or, AST or ALT < 2.5 × ULN (or < 5 × ULN in patients with liver metastases); or, alkaline phosphatase< 2.5 × ULN (or > 5 × ULN in patients with liver metastases,Creatinine clearance > 60 mL/min.
* Signed informed consent.

Exclusion Criteria:

* Prior palliative chemotherapy.
* Received any investigational drug treatment within 30 days of start of study treatment.
* Patients with active gastrointestinal bleeding.
* Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
* History or clinical evidence of brain metastases.
* Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
* Pregnancy women.
* Subjects with reproductive potential not willing to use an effective method of contraception.
* Patients with known active infection with HIV.
* Known hypersensitivity to any of the study drugs.
* Neurological toxicity ≥ grade 2 NCI-CTCAE.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | through study completion, an average of 2 years
  Progression-free survival is determined from the date of treatment to PD or death.

SECONDARY OUTCOMES:
Response rate | up to one year
  the ratio of patients whose efficiency evaluation is CR or PR
Overall survival | OS follow-up period: 18 months or 80% OS events, whichever occurs first.
  the date of treatment to death from any cause or the last follow-up date
Disease control rate | AEs (Adverse events) should be recorded during the study period and six months after last IMP administration
  the ratio of patients whose efficiency evaluation is CR or PR or SD

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D,Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China